CLINICAL TRIAL: NCT07398677
Title: SchoolCare: A Social Intervention Introducing Telepresence Robots and School Navigation to Reduce School Fragmentation for Children Undergoing Cancer Treatment - Study Protocol of a Multi-Site Randomized Controlled Trial (RCT)
Brief Title: SchoolCare: A Social Intervention Introducing Telepresence Robots and School Navigation to Reduce School Fragmentation for Children Undergoing Cancer Treatment
Acronym: SchoolCare
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Hanne Baekgaard Larsen, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: p-2025-19183; 2024-001229 (Other Grant/Funding Number: Danish Childhood Cancer Foundation); 2025-47-1233 (Other Grant/Funding Number: Danish Cancer Research Foundation)
Record Dates: First submitted 2026-01-30; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: School Attendance; Academic Level; Childhood Cancer Survivors; Social Well-being
Keywords: School Attendance; Social well-being; Robot; Telepresence; Cancer; School; Children; School Navigation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Masking Description: The randomization procedure is stratified by site (Copenhagen University Hospital or Aarhus University Hospital/Aalborg University Hospital) and diagnosis (CNS tumor or other cancerous disease). The school navigator and study nurses - responsible for enrolling the children - are blinded to the randomization process. Randomization of the study participants is conducted through REDCap's randomization module, where a random allocation table is generated by a statistician in the research team who, as well as the rest of the research team, is blinded to the randomization table. However, due to the nature of the intervention, neither the research team, school navigator, children nor their parents or teachers are blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Intervention Group (Experimental): Arm A: will in addition to standard care receive a (1) school navigator, (2) a teleteaching program and technical support, and (3) a telepresence robot.
  Interventions: Device: Telepresence robot; Other: School Navigator; Other: Teleteaching and technical support
- Arm B: Comparator group (Active Comparator): Arm B: will in addition to standard care receive a (1) school navigator.
  Interventions: Other: School Navigator

INTERVENTIONS:
Device: Telepresence robot — Children in arm A will receive a telepresence robot (either AV1 or BEAM). In the intervention, children attend their schooling environment through telepresence robots operated via a dedicated application installed on a tablet supplied to each participant. AV1, is a compact unit designed to sit on the student's desk in the classroom. It enables real-time one-way video transmission with zoom functionality combined with two-way audio communication, and allows the user to remotely adjust the robot's orientation, including full rotation and vertical head movement. The second device, BEAM, is a larger, mobile robot positioned on the classroom floor, capable of moving independently within the room at a controlled speed of up to 5 km/h. It offers real-time two-way audio and video interaction via an integrated 10-inch screen with zoom functionality.
  Arms: Arm A: Intervention Group
Other: School Navigator — As part of the SchoolCare intervention, the investigators will hire two professionals with formal education and experience within the school system into roles of school navigators. The primary purpose of the school navigators is to ensure continuous education and to maintain a connection to the schooling environment for children and adolescents diagnosed with cancer. To achieve this, the school navigator will (1) establish contact with the school (teachers and principal) along with the child's first hospital discharge; (2) verify the existence of a learning plan, and if absent, assist the school principal in developing and monitoring an appropriate plan for the child; (3) facilitate ongoing communication with parents through monthly calls throughout the eight-month intervention period; (4) organize a transition meeting at the end of the intervention; and (5) identify barriers and facilitators encountered throughout the intervention period.
Other: Teleteaching and technical support — The school navigator will facilitate a teleteaching program consisting of three components: (1) introduce the robot to parents, school teachers, school principals, and classmates, (2) conduct a teleteaching class where classmates will get hands-on experince with the robot, and (3) provide technical support during the intervention.
  Arms: Arm A: Intervention Group

SUMMARY:
Advances in pediatric cancer treatment have led to markedly improved survival rates, where 5-year survival now exceeds 85%. Despite improved survival, children and adolescents who survive cancer often face significant short- and long-term psychosocial and physical late effects. Children undergoing cancer treatment often experience prolonged school absence, which disrupts academic development and impedes critical socio-emotional growth during formative school years, with lasting consequences into adulthood. Together, these challenges underscore the need for targeted interventions that support educational continuity, promote school activity, and foster psychosocial well-being.

The SchoolCare Intervention aims to reduce school absence experienced by children diagnosed with cancer during their treatment trajectory. The intervention introduces school navigation support in combination with the use of telepresence robots (TPRs) and a teleteaching program. TPRs enables the children to attend school remotely in the classroom when they are not able to attend physically. The study is designed to investigate the effectiveness of the intervention throughout a period of eight months for school-aged children (i.e., 5-17 years) who are diagnosed with cancer. The investigators hypothesize that telepresence robots will increase school attendance among children and adolescents diagnosed with cancer, representing our primary outcome (H1). Additionally, the investigators explore secondary out-comes by hypothesizing that the intervention will improve the social well-being of these children and adolescents (H2) and enhance their academic level (H3). By focusing on both school attendance as well as broader psychosocial and academic effects, this study will provide a comprehensive evaluation of the telepresence robot intervention and its potential to support educational continuity and well-being for children with cancer.

DETAILED DESCRIPTION:
Background: Survival rates for children with cancer have increased substantially. As more children survive their cancer diagnosis, attention has shifted to the educational, social, and psychosocial challenges associated with treatment, including fragmented schooling, social isolation, and risk of long-term academic and social difficulties. Despite legislation ensuring access to education during illness, children often face challenges navigating school, hospital, and home educational systems, highlighting the need for coordinated support. Telepresence robots (TPRs) offer an innovative solution by allowing children to participate remotely in classroom activities while maintaining social presence and inclusion. Although TPRs already have been used for children with medical conditions, no studies have rigorously evaluated their impact on school attendance, social well-being, or academic outcomes for children with cancer. The SchoolCare intervention is a multi-site randomized controlled trial designed to address this gap.

Methods: The SchoolCare intervention is a multi-site, two-arm parallel group (A and B), randomized controlled trial (RCT). The SchoolCare intervention is being conducted at three out of four pediatric oncology treatment centers in Denmark: Copenhagen University Hospital, Aarhus University Hospital, and Aalborg University Hospital. Recruitment will begin in February 2026. After baseline data collection, participants are randomly assigned to either the intervention arm A or B using centrally administered computer-generated random numbers (via R-studio) with a secure, concealed allocation process conducted in REDCap. The randomization procedure is stratified by site (Copenhagen University Hospital or Aarhus University Hospital/Aalborg University Hospital) and diagnosis (CNS tumor or other cancer, or cancer-like, illness). The school navigator and study nurses - responsible for enrolling the children - are blinded to the randomization process, which is conducted by a statistician outside the research team, who is also blinded to baseline data. However, due to the nature of the intervention, neither the research team, school navigator, children nor their parents or teachers are blinded to group assignment.

The intervention comprises three components: (1) a school navigator, (2) a telepresence robot, and (3) a teleteaching program. Participants randomized to Intervention Arm A will receive all three components in addition to standard care. Participants randomized to Intervention Arm B will receive the school navigator component only, in addition to standard care. Two school navigators with professional experience in education will support participants in the SchoolCare intervention-one in the eastern part of Denmark (Copenhagen University hospital) and one in the western part of Denmark (Aarhus and Aalborg University Hospital). Their role is to maintain children's connection to school and ensure continuous learning during treatment. Navigators coordinate between hospital schools, home, and the child's school of origin, supporting learning plans, facilitating communication with parents, and addressing barriers to participation. Monthly calls with parents are conducted for all participants. Navigators receive training on pediatric cancer, the study design, and their responsibilities prior to the intervention.

The two types of telepresence robots are: (1) the AV1, a compact, desk-based robot that supports two-way audio, one-way video streaming with zoom, 360-degree rotation, and head movement, with interactive features such as visual signals and emojis; (2) the BEAM, a larger, floor-based robot that can move around the classroom, offering two-way audio and two-way video streaming on a 10-inch screen with zoom. Participants in intervention arm A will be randomly assigned to receive either an AV1 telepresence robot or a BEAM telepresence robot. Initially, the AV1 is provided for the study participants, until the BEAM is available (expected availability of the BEAM is medio February). Once both types of telepresence robots are available for allocation, the type of telepresence robot provided for each child will alternate between the two types of robots. This means that if the previous child within a distinct randomization group was allocated into arm A and received an AV1 telepresence robot, the next child within that same randomization group, who is allocated into arm A, will receive the BEAM telepresence robot.

The school navigator will lead a teleteaching program with three components: (1) robot introduction, (2) classroom teleteaching, and (3) ongoing technical support. First, the robot will be introduced to the child, parents, and school staff during an initial meeting. Second, the navigator will conduct a teleteaching class in the classroom to familiarize peers and teachers with the robot, drawing on best practices for human-robot interaction and previous studies on telepresence in school settings. Third, the navigator will provide technical support throughout the eight-month intervention period, appoint a key school contact to coordinate communication, and assign one or two classmates as "robot buddies" to support daily robot integration. Patients will be recruited from February 1, 2026, to February 1, 2028, with an expected sample of ~128 children (~64 per intervention arm). Randomization will be 1:1 and stratified by oncology site (Copenhagen vs. Aarhus/Aalborg) and diagnosis (CNS vs. other) to ensure balanced allocation. Accounting for an expected 20% dropout rate, the effective yearly sample is ~64 cases. Sensitivity analyses assume an alpha of 0.05, 95% power, and one primary predictor (school attendance) with five covariates, allowing detection of small-to-medium effect sizes. School attendance will be recorded at monthly intervals through structured telephone calls conducted by the school navigator. The manual registration will be supplemented by school attendance registers. This multi-center randomized controlled trial aims to generate evidence on how telepresence robots can support school participation and reduce educational disruption for children undergoing cancer treatment. By combining remote access to the classroom via telepresence technology with guidance from a school navigator, the study explores innovative approaches to promote both learning continuity and social engagement for affected children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. newly diagnosed with cancer or cancer-like diseases
2. aged 5-17 years
3. admitted to the pediatric oncology ward at Copenhagen University Hospital, Aarhus University Hospital, or Aalborg University Hospital
4. expected to experience disrupted schooling, defined as absence of more than one school day per week over an anticipated period of eight months
5. expected to be enrolled in a school in Denmark during the intervention period

Exclusion Criteria:

1. the children in intervention arm B obtain a telepresence robot outside of the SchoolCare intervention
2. the child is unable to communicate in Danish
3. the child have physical or cognitive impairments that prevent them from operating or meaningfully engaging with the telepresence robot.

Assessment of the latter criterion will be conducted jointly by hospital per-sonnel and the school navigator to determine whether the child is likely to benefit from partic-ipation in the intervention. All reasons for exclusion will be documented and reported.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
School Attendance | From enrollment to the end of treatment at 8 months
  School attendance is measured as the percentage of days attended out of the total number of possible school days. School navigators are instructed to assess school attendance at regular monthly intervals. At each time-point, the school navigator will ask about school attendance during the previous week (at the school of origin, hospital school, or teacher-led homeschooling). If a scheduled monthly assessment coincides with periods when the child is on holiday or hospitalized, the assessment will be conducted during one of the adjacent school weeks (i.e., the week before or the week after). This adjustment applies only if the child misses more than two school days during the assessment week. Holidays and periods of hospitalization are considered legitimate absences and will be accounted for in the calculation of the total number of possible school days. To be included in the analysis, a minimum registration of 25 possible schooldays is required per child.

SECONDARY OUTCOMES:
Social Well-Being | At enrollment, 8 months after inclusion
  Children's social well-being will be assessed using the Danish version of the Strengths and Difficulties Questionnaire (SDQ). The Strengths and Difficulties Questionnaire (SDQ) is a validated tool used to assess social, emotional, and behavioral functioning in children and adolescents. The questionnaire consists of 25 items rated on a three-point scale ranging from "not true" to "certainly true." Responses are grouped into five domains: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. Reporting and scoring will be performed according to the official SDQ guidelines.
Academic Level | At enrollment, 8 months after inclusion
  Children's academic level will be assessed using a 5-point [1; 5] Likert-scale capturing self-reported overall academic performance as well as subject-specific performance in Danish and mathematics. To enhance the validity of the assessment, children's self-reports will be triangulated with corresponding evaluations provided by parents and teachers, allowing for a more comprehensive estimation of the child's academic level. A high value indicates a high academic level, and vice versa.

OTHER OUTCOMES:
School Well-Being | At enrollment, 8 months after inclusion
  School well-being will be measured with questions about school environment, classmates, and teachers (e.g., "Are you [the participants] happy to go to your school?"; "Are you [the participants] happy with your class?"; "Do you [the participants] feel lonely at school?"; "I [the participants] feel that I belong at my school"). The questions all have outcomes within a 5-point Likert scale [1; 5], with total agreement of the statement and total disagreement in each end of the scale.
Self Efficacy | At enrollment, 8 months after inclusion
  Academic self-efficacy. To support the assessment of academic level, children's self-efficacy will be measured using items adapted from the Health Behaviour in School-Aged Children (HBSC) international questionnaire (HBSC International Network, 2023). Two items will be used (i.e., "How often can you [the participants] find a solution to problems in class if you try hard enough?"; "How often can you [the participants] succeed at what you set out to do in class?"). Responses will be recorded according to the HBSC Likert-scale guidelines.
Robot-use | From enrollment to the end of treatment at 8 months
  Datalogs from the telepresence robots will be collected to capture patterns of use, including log-on attempts, session duration, connection failures, and interaction behaviors. This provides insight into how children engage with the technology in real-world school settings. These results will be analyzed exploratory.
Qualitative evaluation of the interventions | 4-8 months after inclusion
  Following the intervention, semi-structured interviews will be conducted with a subset of children diagnosed with cancer, their parents, teachers, and school navigators. The interviews will explore experiences related to school attendance, social well-being, academic level, telepresence robot use, school navigation, and classroom contexts, providing in-depth insights to complement the quantitative outcomes.
  Participant observation will be conducted to explore how the classroom environment and interactions are shaped by the presence of a telepresence robot. The investigators will conduct observations in the classroom settings at the actual schools the children attend.

IPD SHARING:
Plan to Share IPD: Yes
following the final analyses of the study, the IPD will be available upon request
Supporting Information: Study Protocol, SAP